CLINICAL TRIAL: NCT02040948
Title: Accuracy of Pulse Pressure Variation (Nexfin) and of Pleth Variability Index (Radical 7) to Predict the Response to a Fluid Challenge: Comparison With the Reference Method (Measurement of Stroke Volume by Esophageal Doppler)
Brief Title: Accuracy of Pulse Pressure Variation and of Pleth Variability Index to Predict the Response to a Fluid Challenge
Acronym: Nexfin2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011/56; 2011-A01294-37 (Other: ANSM)
Record Dates: First submitted 2014-01-15; First posted 2014-01-20 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Fluid Responsiveness
MeSH Terms: interventions — Stroke Volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical patients (Experimental): * Nexfin (Pulse Pressure Variation)
  * Radical 7 (Pleth Variability Index)
  * CardioQ (stroke volume)
  Interventions: Device: - Nexfin (Pulse Pressure Variation) - Radical 7 (Pleth Variability Index) - CardioQ (stroke volume)

INTERVENTIONS:
Device: - Nexfin (Pulse Pressure Variation) - Radical 7 (Pleth Variability Index) - CardioQ (stroke volume)

SUMMARY:
The aim of this study is to compare the accuracy of Pleth Variability Index (Radical 7 device) and of Pulse Pressure Variation (Nexfin device) with the Doppler measurement of stroke volume (esophageal Doppler) to detect the response to a fluid challenge.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing major abdominal surgical procedures performed by laparotomy
* patients undergoing major urological surgical procedures performed by laparotomy
* patients undergoing major gynecological surgical procedures performed by laparotomy
* age ≥ 18 years
* signed informed consent

Exclusion Criteria:

* pregnant women
* esophageal disease
* aortic valve disease
* allergy to gelatin
* BMI > 35
* beta blocker treatment, antiarrhythmic treatment, arrhythmia, pace-maker,
* presence of an arterio-venous shunt or of any other vascular disease on upper limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Ability of Pleth Variability Index and of Pulse Pressure Variation to detect the response to a fluid challenge | during the intraoperative period
  Three fluid challenges, 250 mL of a gelatine solution, are planned. Pleth Variability Index and Pulse Pressure Variation are compared to the measurement of stroke volume by Esophageal Doppler (the reference method)

SECONDARY OUTCOMES:
Inability to obtain Pleth Variability Index or Pulse Pressure Variation indices | during the intraoperative period

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Beaujon, Clichy, Hauts de Seine
  - Hopital Foch, Suresnes, Hauts de Seine